CLINICAL TRIAL: NCT00527436
Title: Fish Oil and Biomarkers of Cardiovascular Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25918
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Risk Factors
MeSH Terms: interventions — Fish Oils; Fatty Acids, Omega-3; Corn Oil

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Placebo Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Supplement (Other): Fish oil pill
  Interventions: Dietary Supplement: fish oil
- Placebo (Placebo Comparator): Placebo matched corn oil pill
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fish oil — Fish oil pills will be taken daily for 12 weeks
  Other Names: Omega-3 fatty acids
  Arms: Dietary Supplement
Dietary Supplement: Placebo — Placebo (corn oil) will be taken daily for 12 weeks
  Other Names: corn oil
  Arms: Placebo

SUMMARY:
Rationale Experimental data indicate an inverse relation between intake of omega-3 fatty acids ('fish oil'), primarily in the form of eicosapentanoic acid (EPA) and docosahexanoic acid (DHA), and risk of developing cardiovascular disease in healthy adults. Mechanisms underlying this cardioprotective effect are unknown but may involve favorable influences on various biomarkers of cardiovascular risk. In this project we will determine if these favorable effects of omega-3's occur in older healthy adults, as aging is a primary risk factor for cardiovascular disease development.

Key Objectives To determine the effect of chronic (12 week) oral omega-3 fatty acid supplementation on biomarkers of cardiovascular risk in young and older adults. We hypothesize that omega-3 fatty acid supplementation will exert positive effects on biomarkers of cardiovascular risk.

Study Population Healthy young (18-40 years of age) and older (50-79) men and women.

Major Inclusion & Exclusion Criteria Subjects must be healthy (as assessed by history and physical examination: non obese BMI<30: normotensive BP <140/90 mmHg) men and women not currently taking medications that could influence the results. Women must be non-pregnant. Normal liver enzymes (ALT and AST). Individuals with allergies to corn will be excluded.

Allocation to Groups Randomized, double-blinded, and placebo-controlled.

Summary of Procedures Measurements will be made at baseline and repeated ~12 weeks after beginning daily oral ingestion of either low dose or high dose fish oil capsules or placebo

DETAILED DESCRIPTION:
N/A - withdrawn

ELIGIBILITY:
Inclusion Criteria:

Subjects must be healthy (as assessed by history and physical examination:

* Non obese BMI<30: normotensive BP <140/90 mmHg) men and women not currently taking medications that could influence the results.
* Women must be non-pregnant.
* Normal liver enzymes (ALT and AST).

Exclusion Criteria:

* Individuals with allergies to corn will be excluded.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | every 2 weeks for a 12 week duration
  Blood pressure will be measured using a cuff placed around the subject's upper arm as well as a small cuff placed on their finger.
Heart Rate | every two weeks for 12 week duration
  Two-inch square adhesive patches will be used to monitor your heart rate
Arterial Pulse Wave Velocity | every two weeks, for a 12 week duration
  The speed at which blood travels through arteries in the subject's torso will be measured non-invasively using Doppler Flow probes.
Aortic Blood Pressure | every two weeks, for a 12 week duration
  Aortic Blood pressure will be measured non-invasively by pressing an ultrasound probe against an artery in the neck or wrist.
Brachial Artery Blood Flow | every two weeks, for a 12 week duration
  The blood flow into the subject's brachial artery will be measured non-invasively using an ultrasound probe after deflation of a blood pressure cuff that previously had been inflated tightly on the upper forearm for a period of 5 minutes
Brachial Artery Blood flow: After Nitroglycerin (0.4mg) | every two weeks, for a 12 week duration
  The blood flow into the subject's brachial artery will be measured non-invasively using an ultrasound probe after placing a pill containing nitroglycerin (0.4mg) under the tongue.
Microneurography | every two weeks, for a 12 week duration
  Two very fine, sterile nerve wires (micro-electrodes), thinner than a sewing needle, will be introduced through the skin into a nerve located just under the skin of the right leg. This procedure will measure nerve activity from the brain to the leg.

SECONDARY OUTCOMES:
Blood Withdrawal | every two weeks, for a 12 week duration
  An intravenous catheter will be inserted into veins near the elbow to collect blood for standard blood chemistry panel.

OTHER OUTCOMES:
Urine collection | 24 hours
  The subject will be asked to collect urine over the course of one day (24 hours) in a jug provided. The urine will be analyzed for catecholamine levels

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Monahan, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States